CLINICAL TRIAL: NCT02353091
Title: Effects of Remote Microphone Hearing Aids on Classroom Listening, Spatial Listening, and Attention in School-Aged Children With Auditory Processing Disorder
Brief Title: Effects of Remote Microphone Hearing Aids on Children With Auditory Processing Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: GN Resound (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14/0333
Record Dates: First submitted 2015-01-27; First posted 2015-02-02 (Estimated); Results first posted 2020-04-27 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-03

CONDITIONS: Auditory Processing Disorder
MeSH Terms: conditions — Auditory Perceptual Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- APD Control Group (No Intervention): Comprised 13 children diagnosed with APD and acts as a control without using any form of intervention.
- APD Intervention Group (Experimental): Comprised 13 children diagnosed with APD and received the Remote Microphone Hearing AId intervention at the start of the study, after baseline testing, and used for 6 months.
  Interventions: Device: Remote Microphone Hearing Aids

INTERVENTIONS:
Device: Remote Microphone Hearing Aids — The ear receivers connect wirelessly with the microphone being worn by the teacher within a range of 25m.
  Arms: APD Intervention Group

SUMMARY:
Auditory Processing Disorder (APD) is a disorder where the functions of the ear are normal, but the person has difficulty identifying or discriminating sounds and experiences listening difficulties in noise. Remote Microphone Hearing Aids (RMHAs) are wireless listening devices that pick up the speaker's voice and transmit it to a receiver in the listener's ear. In this way, the negative effects of ambient noise, distance from speaker and reverberation are reduced.

The research questions are whether RMHAs improve classroom listening, listening in noise performance, listening in spatialised noise and auditory attention, in children with APD. We hypothesize that RMHA use will lead to improved classroom listening and improved speech-in-noise skills after 6 months of RMHA use. Additionally, we hypothesise that listening in spatialised noise and attention skills will remain unchanged following the intervention period.

Twenty-six (26) children aged 7-12 with a diagnosis of an APD from the Great Ormond Street Hospital Audiology clinic were included in the study.

DETAILED DESCRIPTION:
Auditory Processing Disorder (APD) is a disorder where the functions of the ear (outer, middle, inner) are normal but the person has difficulty identifying or discriminating sounds (1). For children with APD it is particularly difficult to hear when the listening conditions are not ideal. For example, when there is background noise it becomes really challenging to focus on the speaker. Two other factors that influence their hearing ability are reverberation and the distance from the speaker (2). Some symptoms reported for APD are listening difficulties in background noise, attention and memory problems, and distractibility (3,4). Children with APD have worse skills in speech perception in noise compared to typically developing children (5,6) and have also have poorer sustained auditory attention compared to children suspected of APD (7).

Remote Microphone Hearing Aids (RMHAs) are a management approach recommended for children with APD. These are wireless listening devices that pick up the speaker's voice and transmit it to a receiver in the listener's ear. The use of this system helps improve the signal-to-noise ratio for children and bypasses the negative effects of background noise and reverberation in the classroom (2,8,9). There have not been many studies, though. That looked into the effects of RMHA on children with APD. Previous research suggests that children with APD after a prolonged use of RMHAs benefit from improved speech perception which is possibly linked to an enhanced auditory system (9). Adding to that, children with APD have shown improved speech in noise perception when using the RMHA, hence emphasizing the advantages of the device in discriminating speech in background noise (9,10).

Sustained attention and the ability of children with APD to listen in spatialised noise after RMHA use has been examined by one study (10). It did not show improvement (unaided) in any of the two tests. However, this was a non-randomised trial that did not use a control group. As the central point of this study will be the use of the RMHA by children with APD for 6 months, it is expected that the findings could add valuable information on the subject.

Aim and hypotheses The aim of the study is to examine the effect of a 6-month RMHA use on self-reported listening in the classroom, speech perception in noise, speech perception in spatialised noise and on attention skills.

Hypotheses:

i. Children with APD who use RMHAs will show greater improvements in classroom listening, listening in noise and sustained auditory attention (unaided) after 6 months of RMHA use in comparison to the APD control group.

ii. Children with APD who use the RMHA will not show greater improvements in listening in spatialised speech noise and divided and visual attention measures after 6 months of RMHA use in comparison to the APD control group.

Research Design and Methodology Participants and Recruitment We recruited 26 children aged 7-12 years. All children have been diagnosed and referred from the Auditory Processing Disorders Clinic at Great Ormond Street Hospital. The total sample size was decided using this power sample: N = 24 (total sample size) calculated using the F test for repeated measures between-within interaction ANOVA based on an estimated 0.5 effect size f(U), 80% power, at 5% significance, using 2 groups and 3 measurement points. Accounting for a 10% loss due to follow-up, the final study sample size comprised 26 children.

Inclusion criteria:

1. Diagnosis of APD based on clinical tests administered by qualified audiologists as per the clinic's diagnosis protocol.
2. No neurological or pervasive disorder or developmental delay (e.g. Attention Deficit Hyperactivity Disorder, epilepsy, Autism Spectrum Disorder, Developmental Language Disorder, Down Syndrome).
3. Non-verbal cognitive ability score of 85 or greater.
4. Ages between 7-12 years.
5. Native English speakers.
6. No prior use of RMHAs. Subjects were semi-randomly assigned to each of two intervention arms. The two groups were stratified for age and balanced for gender.

Children were given RMHAs to use at school and were compared to the control that did not use any intervention for the study period. Children were enrolled in the study for 6 months. All groups were tested before the start of the RMHA intervention, after 3 months, and at the end of the study (after 6 months).

Explanation of each test:

1. A hearing test (Pure Tone Audiometry approx. 10mins). To determine their hearing is normal.
2. Non-verbal IQ test (Weschler test of non-verbal intelligence). To be performed by the PhD Student. (approx. 15mins). To assess determine whether their intelligence level is above normal.
3. Listening in spatialised noise test (LiSN-S, approx. 15mins). To be administered through the use of headphones by the PhD student. To determine their listening in spatialised speech noise abilities.
4. The Test of Everyday Attention for Children (TEACh). To be conducted as play type activities by the PhD student after receiving sufficient training by the clinical psychologist. (approx. 45mins possibly cut down to 30mins). To assess their attention.
5. Two questionnaires to be filled by the children's parents.

   1. The Children's Communication Checklist-2 (CCC-2). A 70-item questionnaire which screens for communication problems (including language disorders and autism).
   2. The Children's Auditory Performance Scale (CHAPS). It assesses aspects of children's listening.
6. One questionnaire to be completed by the children (Listening Inventory For Education-Revised [LIFE-R] for assessing their listening difficulty.

Data analysis:

Data were analysed in SPSS statistics software, using mixed ANOVA. Group was the between-subjects factor and time was the within-subjects factor.

Ethical issues

School and teacher involvement:

The teachers of the children who received the RMHA were provided with an information sheet and consent form and were required to wear the microphone (which picks up the teacher's voice and transmits it wirelessly to the ear receivers in the child's ear) for the duration of lecture-based subjects. Remote microphone hearing aids are generally beingg provided (funded by the school budget) to some children after clinical recommendations and this is not an unusual situation within the school environment.

We liaised with the teacher of the school to ensure that the school was aware that the student has been issued with the RMHA. A general guide for the system was made available in addition to information conveyed by the PhD student.

Informed consent:

The child's parents were given detailed written information and consent forms to sign. They were given up to a week to study and decide whether they wished for their child to participate in the study. They were only allowed to take part once they have understood the purpose and procedures of the study and they signed the consent forms. In addition, children were also given information sheets adjusted to their age. Written assent from children in the presence of their parents or carers was sought.

Rights to withdraw from the study:

This was outlined on both the information sheet and consent form and explained verbally during test visits. This information stated that participants were allowed to withdraw from the study at any point should they wished to. Withdrawal from the study did not involve any penalty or loss of benefit to them - this information was clearly underlined at the information sheet and verbally communicated.

Data protection:

Parents of the participants and the participants were informed that their information was anonymised and kept confidential. Data was anonymised prior to analysis by the use of participant codes. Storage of the data was in accordance with the data protection act 1998.

Other issues:

None of these tests were invasive or unpleasant, and they were conducted in comfortable sound levels (slightly higher than the usual conversational level).

References

1. Dawes P, Bishop DVM. Auditory Processing Disorder in Relation to Developmental Disorders of Language, Communication and Attention: A Review and Critique. Int J Lang Commun Disord [Internet]. 2009 [cited 2014 Apr 1];44(4):440-65. Available from: http://www.ncbi.nlm.nih.gov/pubmed/19925352
2. Keith WJ, Purdy SC. Assistive and Therapeutic Effects of Amplification for Auditory Processing Disorder. Semin Hear [Internet]. 2014;35(1):27-38. Available from: https://www.thieme-connect.com/products/ejournals/html/10.1055/s-0033-1363522
3. American Speech-Language-Hearing Association. (Central) Auditory Processing Disorders. Technical Report [Internet]. American Speech-Language-Hearing Association. 2005 [cited 2019 Aug 6]. Available from: http://www.asha.org/policy/TR2005-00043/
4. American Academy of Audiology. American Academy of Audiology Clinical Practice Guidelines. Diagnosis, Treatment and Management of Children and Adults with Central Auditory Processing Disorder [Internet]. American Academy of Audiology. 2010 [cited 2019 Aug 6]. p. 1-51. Available from: http://www.audiology.org/publications-resources/document-library/central-auditory-processing-disorder
5. Lagacé J, Jutras B, Giguère C, Gagné J-P. Speech Perception in Noise: Exploring the Effect of Linguistic Context in Children With and Without Auditory Processing Disorder. Int J Audiol [Internet]. 2011;50(6):385-95. Available from: https://www.ncbi.nlm.nih.gov/pubmed/21599614
6. Rocha-Muniz CN, Zachi EC, Teixeira RAA, Ventura DF, Befi-Lopes DM, Schochat E. Association Between Language Development and Auditory Processing Disorders. Braz J Otorhinolaryngol [Internet]. 2014;80(3):231-6. Available from: http://www.ncbi.nlm.nih.gov/pubmed/25153108
7. Allen P, Allan C. Auditory Processing Disorders: Relationship to Cognitive Processes and Underlying Auditory Neural Integrity. Int J Pediatr Otorhinolaryngol [Internet]. 2014;78(2):198-208. Available from: http://dx.doi.org/10.1016/j.ijporl.2013.10.048
8. British Society of Audiology. Practice Guidance. An Overview of Current Management of Auditory Processing Disorder (APD) [Internet]. British Society of Audiology. 2011 [cited 2019 Aug 6]. p. 1-60. Available from: http://www.thebsa.org.uk/docs/docsfromold/BSA_APD_Management_1Aug11_FINAL_amended17Oct11.pdf
9. Johnston KN, John AB, Kreisman N V, Hall III JW, Crandell CC. Multiple Benefits of Personal FM System use by Children with Auditory Processing Disorder (APD). Int J Audiol [Internet]. 2009 Jan;48(6):371-83. Available from: http://www.ncbi.nlm.nih.gov/pubmed/19925345
10. Smart JL, Purdy SC, Kelly AS. Impact of Personal Frequency Modulation Systems on Behavioral and Cortical Auditory Evoked Potential Measures of Auditory Processing and Classroom Listening in School-Aged Children with Auditory Processing Disorder. J Am Acad Audiol [Internet]. 2018;19:1-19. Available from: http://www.ingentaconnect.com/content/10.3766/jaaa.16074

ELIGIBILITY:
Inclusion criteria:

1. Normal audiogram.
2. Diagnosis of APD based on clinical tests administered by qualified audiologists as per the clinic's diagnosis protocol.
3. No neurological or pervasive disorder or developmental delay (e.g. Attention Deficit Hyperactivity Disorder, epilepsy, Autism Spectrum Disorder, Developmental Language Disorder, Down Syndrome).
4. Non-verbal cognitive ability score of 85 or greater.
5. Ages between 7-12 years.
6. Native English speakers.
7. No prior use of RMHAs.

Exclusion criteria:

Any violation of the above conditions.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doris-Eva Bamiou, MD MSc PhD, Principal Investigator — UCL Ear Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dawes P, Bishop D. Auditory processing disorder in relation to developmental disorders of language, communication and attention: a review and critique. Int J Lang Commun Disord. 2009 Jul-Aug;44(4):440-65. doi: 10.1080/13682820902929073. PMID 19925352
- [Background] Lagace J, Jutras B, Giguere C, Gagne JP. Speech perception in noise: exploring the effect of linguistic context in children with and without auditory processing disorder. Int J Audiol. 2011 Jun;50(6):385-95. doi: 10.3109/14992027.2011.553204. PMID 21599614
- [Background] Rocha-Muniz CN, Zachi EC, Teixeira RA, Ventura DF, Befi-Lopes DM, Schochat E. Association between language development and auditory processing disorders. Braz J Otorhinolaryngol. 2014 May-Jun;80(3):231-6. doi: 10.1016/j.bjorl.2014.01.002. PMID 25153108
- [Background] Allen P, Allan C. Auditory processing disorders: relationship to cognitive processes and underlying auditory neural integrity. Int J Pediatr Otorhinolaryngol. 2014 Feb;78(2):198-208. doi: 10.1016/j.ijporl.2013.10.048. Epub 2013 Nov 20. PMID 24370466
- [Background] Johnston KN, John AB, Kreisman NV, Hall JW 3rd, Crandell CC. Multiple benefits of personal FM system use by children with auditory processing disorder (APD). Int J Audiol. 2009;48(6):371-83. doi: 10.1080/14992020802687516. PMID 19925345
- [Background] Smart JL, Purdy SC, Kelly AS. Impact of Personal Frequency Modulation Systems on Behavioral and Cortical Auditory Evoked Potential Measures of Auditory Processing and Classroom Listening in School-Aged Children with Auditory Processing Disorder. J Am Acad Audiol. 2018 Jul/Aug;29(7):568-586. doi: 10.3766/jaaa.16074. PMID 29988006
- [Derived] Stavrinos G, Iliadou VV, Pavlou M, Bamiou DE. Remote Microphone Hearing Aid Use Improves Classroom Listening, Without Adverse Effects on Spatial Listening and Attention Skills, in Children With Auditory Processing Disorder: A Randomised Controlled Trial. Front Neurosci. 2020 Aug 21;14:904. doi: 10.3389/fnins.2020.00904. eCollection 2020. PMID 32973443

RESULTS

PARTICIPANT FLOW:
Groups:
- APD Control Group: Comprised 13 children diagnosed with APD and did not receive an intervention.
- APD Intervention Group: Comprised 13 children diagnosed with APD and received the Remote Microphone Hearing Aid intervention right after baseline and for 6 months.
Period: Overall Study
Arm/Group | APD Control Group | APD Intervention Group
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- APD Control Group: Comprised 13 children diagnosed with APD and rdid not receive an intervention.
- Total: Total of all reporting groups
Arm/Group | APD Control Group | APD Intervention Group | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: Months] | 116 (16.3) | 115 (16.1) | 115 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 9 | 9 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Listening Inventory For Education Revised (LIFE-R) - Total Score
Description: Children questionnaire measured in raw scores. This is the total score of 9 questions on a likert scale from 0 to 5. Thus, this is the summed score. Therefore, minimum value 0, maximum value 45. Higher scores mean better outcome.
Time Frame: Baseline to 6 months
Population: An outlier at the 3-month time-point (at -3.25 SDs) was removed
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- APD Control Group: Comprised of 13 children diagnosed with APD and does not receive any intervention.
Arm/Group | APD Control Group | APD Intervention Group
Number analyzed (Participants) | 12 | 13
Units on a scale
  Baseline | 30.91 (4.46) | 28.30 (7.44)
  3 months | 33.33 (5.59) | 35.61 (3.45)
  6 months | 30.83 (5.06) | 33.30 (7.66)

2. Primary Outcome: Listening in Spatialised Noise - Sentences Test (LiSN-S) - Low-cue Speech Reception Threshold Condition
Description: Speech in noise test measured in z scores. Minimum value -2, maximum value +2. Higher scores mean better outcome. Z scores are automatically calculated in the computer test software based on normative sample data on decibel (dB) measures.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Error); unit: z scores
Arm/Group | APD Control Group | APD Intervention Group
Number analyzed (Participants) | 13 | 13
z scores
  Baseline | -0.56 (0.90) | -0.99 (1.12)
  3 months | -0.46 (1.43) | -0.63 (1.61)
  6 months | -1.38 (3.33) | -1.05 (1.51)

3. Primary Outcome: Listening in Spatialised Noise - Sentences Test (LiSN-S) - High-cue Speech Reception Threshold Condition
Description: as for outcome 2
Time Frame: 6 months
Population: One outlier in the intervention group was found. Outlier was removed as participant had decreased focus and difficulty remaining seated during this condition.
Measure: Mean (Standard Deviation); unit: z scores
Groups:
- APD Control Group: Comprised of 13 children diagnosed with APD and did not receive any intervention.
Arm/Group | APD Control Group | APD Intervention Group
Number analyzed (Participants) | 13 | 12
z scores
  Baseline | -0.83 (1.45) | -1.27 (1.02)
  3 months | -0.70 (1.34) | -0.60 (1.08)
  6 months | -1.23 (1.82) | -0.68 (1.66)

4. Primary Outcome: Listening in Spatialised Noise - Sentences Test (LiSN-S) - Talker Advantage Condition
Description: as for outcome 2
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: z scores
Arm/Group | APD Control Group | APD Intervention Group
Number analyzed (Participants) | 13 | 13
z scores
  Baseline | -1.01 (1.14) | -0.84 (0.80)
  3 months | -0.32 (1.00) | -0.59 (0.82)
  6 months | -0.44 (1.11) | -0.68 (0.93)

5. Primary Outcome: Listening in Spatialised Noise - Sentences Test (LiSN-S) - Spatial Advantage Condition
Description: as for outcome 2
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: z scores
Arm/Group | APD Control Group | APD Intervention Group
Number analyzed (Participants) | 13 | 13
z scores
  Baseline | -1.50 (1.54) | -0.97 (1.07)
  3 months | -1.31 (1.41) | -0.99 (1.57)
  6 months | -0.98 (1.76) | -0.53 (1.35)

6. Primary Outcome: Listening in Spatialised Noise - Sentences Test (LiSN-S) - Total Advantage Condition
Description: as for outcome 2
Time Frame: Baseline to 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: z scores
Arm/Group | APD Control Group | APD Intervention Group
Number analyzed (Participants) | 13 | 12
z scores
  Baseline | -0.56 (1.34) | -0.94 (1.12)
  3 months | -0.52 (1.28) | -0.47 (1.06)
  6 months | -0.63 (1.07) | -0.30 (1.28)

7. Secondary Outcome: Test of Everyday Attention for Children TEACh - Sustained Auditory Attention Subscale
Description: A validated attention test to test children's auditory attention. Measured on scaled scores. Minimum value 1, maximum value 19. Higher scores mean better outcome.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: scaled scores
Groups:
- APD Control Group: Comprised 13 children diagnosed with APD and did not receive any intervention.
- APD Intervention Group: Comprised 13 children diagnosed with APD and received a Remotre Microphone Hearing Aid intervention after baseline testing and for 6 months.
Arm/Group | APD Control Group | APD Intervention Group
Number analyzed (Participants) | 13 | 13
scaled scores
  Baseline | 9.76 (4.00) | 6.30 (2.62)
  3 months | 7.76 (3.67) | 6.61 (3.84)
  6 months | 8.23 (4.22) | 5.76 (1.87)

8. Secondary Outcome: Test of Everyday Attention for Children TEACh - Divided Auditory-Visual Attention Subscale
Description: A validated attention test to test children's auditory-visual attention. Measured on scaled scores. Minimum value 1, maximum value 19. Higher scores mean better outcome.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: scaled scores
Arm/Group | APD Control Group | APD Intervention Group
Number analyzed (Participants) | 13 | 13
scaled scores
  Baseline | 6.61 (3.17) | 2.38 (2.39)
  3 months | 5.23 (2.83) | 5.15 (3.67)
  6 months | 5.92 (3.25) | 5.76 (2.16)

9. Secondary Outcome: Test of Everyday Attention for Children TEACh - Selective Visual Attention Subscale
Description: A validated attention test to test children's visual attention. Measured on scaled scores. Minimum value 1, maximum value 19. Higher scores mean better outcome.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: scaled scores
Arm/Group | APD Control Group | APD Intervention Group
Number analyzed (Participants) | 13 | 13
scaled scores
  Baseline | 9.69 (2.01) | 6.00 (2.85)
  3 months | 10.30 (3.61) | 8.30 (2.71)
  6 months | 10.92 (1.93) | 9.61 (2.32)

10. Secondary Outcome: Test of Everyday Attention for Children TEACh - Divided Auditory Attention Subscale
Description: as for outcome 7
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: scaled scores
Arm/Group | APD Control Group | APD Intervention Group
Number analyzed (Participants) | 13 | 13
scaled scores
  Baseline | 9.15 (3.13) | 6.53 (3.12)
  3 months | 8.61 (4.21) | 6.76 (2.55)
  6 months | 8.69 (4.17) | 6.07 (3.17)

11. Other Pre Specified Outcome: Children's Auditory Performance Scale - Noise Subscale
Description: Parental questionnaire measured in raw unstandardised scores. Minimum value is -5, maximum value is +1. Higher score means better outcome.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- APD Control Group: Comprised 13 children diagnosed with APD that did not receive any intervention.
- APD Intervention Group: Comprised 13 children diagnosed with APD that received the Remote Microphone Hearing Aid intervention after baseline testing and used for 6 months.
Arm/Group | APD Control Group | APD Intervention Group
Number analyzed (Participants) | 13 | 13
units on a scale
  Baseline | -2.85 (1.01) | -3.29 (0.89)
  3 months | -2.36 (1.31) | -2.82 (0.83)
  6 months | -2.19 (1.07) | -2.95 (0.97)

12. Other Pre Specified Outcome: Children's Auditory Performance Scale - Multiple Inputs Subscale
Description: as for outcome 11
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | APD Control Group | APD Intervention Group
Number analyzed (Participants) | 13 | 13
Units on a scale
  Baseline | -1.31 (0.99) | -1.62 (1.21)
  3 months | -1.33 (1.09) | -1.21 (1.00)
  6 months | -1.05 (1.14) | -1.33 (1.41)

13. Other Pre Specified Outcome: Children's Auditory Performance Scale - Auditory Memory Sequencing Subscale
Description: as for outcome 11
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | APD Control Group | APD Intervention Group
Number analyzed (Participants) | 13 | 13
Units on a scale
  Baseline | -1.77 (1.15) | -2.63 (1.53)
  3 months | -2.24 (1.30) | -2.06 (1.33)
  6 months | -2.14 (1.35) | -2.51 (1.41)

14. Other Pre Specified Outcome: Children's Auditory Performance Scale - Auditory Attention Span Subscale
Description: as for outcome 11
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | APD Control Group | APD Intervention Group
Number analyzed (Participants) | 13 | 13
Units on a scale
  Baseline | -1.34 (0.86) | -1.84 (1.16)
  3 months | -1.62 (1.06) | -1.57 (0.93)
  6 months | -1.46 (1.04) | -1.77 (1.17)

15. Other Pre Specified Outcome: The Children's Communication Checklist - 2 - Standard Language Composite Score
Description: Parental questionnaire. Average composite of scaled scores are used to calculate the outcome, so units are scaled scores. Maximum value is 1, maximum value is 19. Higher score means better outcome.
Time Frame: 6 months
Population: One parent from intervention group did not complete any of the questionnaires, hence intervention group number analysed was 12.
Measure: Mean (Standard Deviation); unit: scaled scores
Groups:
- APD Group 1: APD Group 1 is comprised of 13 children diagnosed with APD and receives the device from the beginning of the study.
  Personal FM system
- APD Group 2: APD Group 2 is comprised of 13 children diagnosed with APD and receives the device 6 months later than APD Group 1.
  Personal FM system
Arm/Group | APD Group 1 | APD Group 2
Number analyzed (Participants) | 13 | 12
scaled scores
  Baseline | 5.82 (2.65) | 5.44 (2.56)
  3 months | 6.03 (2.71) | 5.39 (2.88)
  6 months | 6.50 (2.84) | 5.58 (2.35)

16. Other Pre Specified Outcome: The Children's Communication Checklist - 2 - Non-Standard Language Composite Score
Description: as for outcome 15
Time Frame: Baseline to 6 months
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: scaled scores
Arm/Group | APD Control Group | APD Intervention Group
Number analyzed (Participants) | 13 | 12
scaled scores
  Baseline | 6.25 (2.82) | 6.19 (2.66)
  3 months | 6.38 (2.87) | 6.08 (2.60)
  6 months | 6.61 (3.06) | 5.70 (2.83)

17. Other Pre Specified Outcome: Screening Instrument For Targeting Educational Risk Performance Scale - Attention Subscale
Description: Raw unstandardised score measured in Likert Scale (5 scales). Minimum score is 1, maximum score is 5. Higher score means better outcome. The three Attention Subscales are averaged to create one combined score.
Time Frame: 6 months
Population: Only 5 questionnaires given to teachers were returned, all from the intervention group. The data for these 5 questionnaires are presented in the APD Group 2, as all 5 cases are from that group only. Group 1 has no data.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- APD Group 1: APD Group 1 is comprised 13 children diagnosed with APD and acts as a control without using any form of intervention.
  No intervention: No intervention is assigned
- APD Group 2: APD Group 2 is comprised 13 children diagnosed with APD and receives the intervention at the start of the study.
  Remote Microphone Hearing Aids: The ear receivers connect wirelessly with the microphone being worn by the teacher within a range of 25m.
Arm/Group | APD Group 1 | APD Group 2
Number analyzed (Participants) | 0 | 5
units on a scale
  Baseline |  | 2.33 (0.59)
  6 months |  | 2.79 (1.00)

ADVERSE EVENTS:
Time Frame: Adverse event data were collection for a period of 6 months.
Description: The concern that spatial listening of children would be affected by the intervention was monitored through the use of the Listening in Spatialised Noise - Sentences test.
Arm/Group | APD Control Group | APD Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

LIMITATIONS AND CAVEATS:
Placebo, Hawthorne or observer bias effects may have influenced the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2015-09-29): https://cdn.clinicaltrials.gov/large-docs/91/NCT02353091/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/91/NCT02353091/Prot_SAP_001.pdf